CLINICAL TRIAL: NCT04208022
Title: The Effect of Hypermobility on Respiratory Functions in Musicians Playing Wind Instruments and Healthy Individuals Not Involved in Music
Brief Title: The Effect of Hypermobility Healthy Individuals
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istanbul Kültür University (Other)
Collaborators: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Gülşah Karaca, Research Assistant, Istanbul Kültür University
Other Study IDs: IstanbulKulturU
Record Dates: First submitted 2019-12-16; First posted 2019-12-23 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Respiratory Problems
Keywords: Musicians; Respiratory; Hypermobility

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy Musician: At least 15 hypermobile musicians and at least 15 non-hypermobile musicians will be included in the study.
  Interventions: Other: Respiratory evaluation
- Healthy Individuals: The study will include at least 15 healthy non-hypermobile individuals who do not deal with music and at least 15 healthy hypermobile individuals who do not deal with music.
  Interventions: Other: Respiratory evaluation

INTERVENTIONS:
Other: Respiratory evaluation — Hypermobility and Respiratory evaluation

SUMMARY:
Benign Joint Hypermobility Syndrome is a hereditary connective tissue problem characterized by the emergence of multiple musculoskeletal problems in hypermobile individuals without a systemic rheumatologic disease. Studies have shown that hypermobility may also affect lung function. Playing wind instruments requires tiring breathing activity. The effect of wind instrument on lung function and how it affects lung function is a highly controversial issue. Given the distribution and importance of collagen tissue in the body, multiple effects of hypermobility are inevitable. The aim of this study was to evaluate the presence of hypermobility in young healthy individuals; The aim of the study is to investigate the effects of hypermobility on the cardiovascular system and to provide training to the participants regarding the findings.The aim of this study is to investigate the relationship of hypermobility with respiratory functions in professional hypermobile musicians and to compare this relationship with healthy hypermobile individuals who are not engaged in music.

DETAILED DESCRIPTION:
Sociodemographic data and musical backgrounds of all cases will be recorded. In accordance with the objectives, erm Upper Extremity Hypermobility Assessment Questionnaire "was used for hypermobility, pulmonary function test, respiratory and oral pressure measurement and respiratory muscle strength. The George Respiratory Questionnaire (SGRQ) will be used to assess the quality of life associated with respiration and the risk of asthma with the ile European Respiratory Health Survey, Phase 1 "questionnaire.We believe that the effects of hypermobility on pulmonary functions in healthy individuals will be clarified if this study takes place.

ELIGIBILITY:
Inclusion Criteria for Musicians

Be between 18-35 years Playing wind instruments for at least one year For the hypermobile subgroup; Obtaining ≥7 / 12 points from the Upper Extremity Hypermobility Assessment Questionnaire

Inclusion Criteria for Healthy Individuals Not Engaged in Music

Be between 18-35 years No diagnosed health problems For the hypermobile subgroup; Obtaining ≥7 / 12 points from the Upper Extremity Hypermobility Assessment Questionnaire

Exclusion Criteria for Musicians

Having a specific respiratory problem diagnosed Symptoms of nerve impingement in upper extremity Smoking

Exclusion Criteria for Healthy Individuals Not Engaged in Music

Symptoms of nerve impingement in upper extremity Smoking

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The musicians who meet the criteria for inclusion in the study and who play the wind instrument who agree to voluntarily participate in the study and healthy individuals who are not interested in music will be included.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
The Upper Limb Hypermobility Assessment Tool | 10 minutes
  Hypermobility
St. George Respiratory Questionnaire | 5 minutes
  respiratory quality
European Respiratory Health Survey, Phase 1 | 5 minutes
  assess the risk of asthma
Respiratory function test | 15minutes
  FEV1,FVC
mouth pressure measurement | 15minutes
  MIP, MEP

SECONDARY OUTCOMES:
Musculoskeletal Pain Intensity and Interference Questionnaire for Musicians | 10 minutes
  Pain

CONTACTS AND LOCATIONS:
Overall Officials: Esra Pehlivan, Asst.Prof.Dr, Principal Investigator — Saglik Bilimleri Universitesi; Gulsah Karaca, Researcher, Principal Investigator — Istanbul Kültür University
Locations (1):
- Istanbul Kultur University, Istanbul, E5 Highway Bakırköy, İstanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided